CLINICAL TRIAL: NCT01493401
Title: Exploration of the Potential of Urinary Nerve Growth Factor (NGF) as a Biomarker for Diagnosis and Prognosis of Mixed Urinary Incontinence After Midurethral Slings
Brief Title: Urinary Urinary Nerve Growth Factor (NGF) as a Biomarker for Mixed Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Urology, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009-11-068
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Mixed Urinary Incontinence
MeSH Terms: interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midurethral sling (Experimental): Currently available midurethral procedures for stress urinary incontinence can be used.
  Interventions: Procedure: Midurethral slings (MUS)

INTERVENTIONS:
Procedure: Midurethral slings (MUS) — Retropubic, Transobturator, and Single incision MUS can be used.
  Other Names: TVT, TVT-O, TOT, TVT-Secur, Needleless, etc.

SUMMARY:
Female urinary incontinence (UI) can be caused by pure stress UI (SUI), pure urgency UI (UUI) and mixed SUI and UUI (MUI). Clinically it might not be that easy to separate MUI and SUI. Patients might perceive urgency when they have an incompetent urethra and a full bladder.

Urinary tract nerve growth factor (NGF)is produced by bladder urothelium and smooth muscle. Increased levels of NGF have been reported in the bladder tissue and urine of patients with overactive bladder (OAB).

If the urinary levels of NGF differ among women with pure SUI and MUI, then urinary NGF level might be a biomarker in the differential diagnosis of MUI in women.

Also, decreased urinary NGF level was reported in OAB patients of whom the symptoms were improved. So, we might expect that the remnant OAB symptom including urgency incontinence can be improved, if the urinary NGF levels decrease after midurethral slings for SUI in MUI patients.

We aimed to explore the value of the urinary NGF as a biomarker for differential diagnosis and as a prognostic marker for predicting the improvement of OAB symptom after midurethral slings.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or over 18 years with MUI for 3 or over 3 months
* Proven SUI by urodynamic study (UDS)or stress test
* Abdominal leak point pressure (ALPP)of 120 or less than 120cmH2O in UDS
* Symptoms verified using 5 day bladder diary as below i) number of urgency incontinence; 3 or more than 3/5days ii) number of micturition; 8 or more than 8/24hrs iii) number of urgency; 2 or more than 2/24hrs
* Women who cannot be pregnant or do not have plan to be pregnant
* Ability and willingness to correctly complete the micturition diary and questionnaire
* Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

* The subject has WBC≧3, Albumin≧+1, Nit ≧+1 upon urinalysis
* On an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
* Patient has a significant pelvic orgen prolapse (POP) of ICS Stage 3 or over 3.
* Patients with combined POP surgery.
* Patients with bladder outlet obstruction on UDS or physical exam
* Patients with detrusor underactivity
* Diagnosed or suspected interstitial cystitis or bladder cancer
* History of radiation therapy on pelvic cavity
* Patients with neurologic condition which can affect lower urinary tract function
* History of urogenical malignancy within recent 2 years
* Treatment within the 14 days preceding enrollment, or expected to initiate treatment during the study with:

  i)Any anticholinergic drugs and any drug treatment affecting lower urinary tract function Estrogen treatment started more than 2 months prior to inclusion is allowed. ii) electrostimulation, bladder training, electromagnetic treatment
* Patient is on anti-coagulation therapy.
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Difference in the baseline urinary NGF level between patients with and without urgency incontinence at 6 months after midurethral slings | 6 months after midurethral slings

SECONDARY OUTCOMES:
Baselinec cut-off value of urinary NGF level which can predict the patients whose urgency incontinence will be cured and whose urgency incontinence will not be cured. | 6 months after midurethral slings
Difference in urinary NGF level between pure SUI and MUI patients | Baseline
Changes in OAB symptoms (including urgency incontinence) and SUI after midurethral slings | 2 and 6 months after midurethral slings
Correlation between changes in urinary NGF and OAB symptoms (including urgency incontinence) after midurethral slings | 2 and 6 months after midurethral slings

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - The Catholic University of Korea College of Medicine, Bucheon St. Mary's Hospital, Bucheon-si
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul